CLINICAL TRIAL: NCT00636987
Title: Post-Approval Study Protocol of the St. Jude Medical Biocor and Biocor Supra Valves
Brief Title: Aortic or Mitral Valve Replacement With the Biocor and Biocor Supra
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0505
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Aortic Valve Insufficiency; Aortic Valve Regurgitation; Aortic Valve Stenosis; Aortic Valve Incompetence; Mitral Valve Insufficiency; Mitral Valve Regurgitation; Mitral Valve Stenosis; Mitral Valve Incompetence
Keywords: aortic valve; mitral valve; heart valve; tissue valve; bioprosthesis; valve disorder; valve disease; cardiac surgery; aortic valve regurgitation; aortic valve stenosis; mitral valve regurgitation; mitral valve stenosis
MeSH Terms: conditions — Aortic Valve Insufficiency; Aortic Valve Stenosis; Mitral Valve Insufficiency; Mitral Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Implanted with Biocor or Biocor Supra Valves (Other)
  Interventions: Device: Biocor and Biocor Supra valves

INTERVENTIONS:
Device: Biocor and Biocor Supra valves — Replacement for a diseased, damaged, malformed aortic or mitral heart valve
  Other Names: Heart Valve Replacement

SUMMARY:
The purpose of this study is to further evaluate the long-term safety and effectiveness of the Biocor and Biocor Supra Valves.

DETAILED DESCRIPTION:
The clinical investigation is a multi-center, prospective, non-randomized, observational, FDA-required post-approval study designed to further evaluate the safety and effectiveness of the Biocor and Biocor Supra Valves.

ELIGIBILITY:
Inclusion Criteria:

* Requires aortic or mitral valve replacement (heart surgery such as bypass is allowed at the same time)
* Legal age
* Signed informed consent prior to surgery
* Willing to complete all follow-up requirements

Exclusion Criteria:

* Pregnant or nursing women
* Already have had a valve replaced other than that for the scheduled replacement
* Needs another valve replaced
* Cannot return for required follow-up visits
* Have active endocarditis
* Acute preoperative neurological event (such as a stroke)
* Renal dialysis
* History of substance abuse within one year or is a prison inmate
* Participating in another study
* Had the Biocor or Biocor Supra valve implanted but then the device was explanted
* Life expectancy less than five years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2007-04; Primary Completion 2015-10 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Urban Lonn, MD, PhD, Study Director — Abbott Medical Devices
Locations (17):
- United States (17):
  - Scripps Green Hospital/Scripps Clinic, La Jolla, California
  - USC University Hospital, Department of Cardiothoracic Surgery, Los Angeles, California
  - The Heart Group, PC, Evansville, Indiana
  - Indiana Heart Hospital, Indianapolis, Indiana
  - Maine Medical Center, Portland, Maine
  - HealthEast St. Joseph Hospital, Saint Paul, Minnesota
  - St. Luke's Hospital, Kansas City, Missouri
  - Catholic Medical Center, Manchester, New Hampshire
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Saint Thomas Hospital, Nashville, Tennessee
  - Sentara Norfolk General Hospital/Sentara Heart Hospital, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Implanted With Biocor or Biocor Supra Valves
Started | 297
Completed | 108
Not Completed | 189
Not completed — Death | 44
Not completed — Explanted | 13
Not completed — Lost to Follow-up | 63
Not completed — 5 year visit window not complete | 69

BASELINE CHARACTERISTICS:
Arm/Group | Implanted With Biocor or Biocor Supra Valves
Number analyzed (Participants) | 297
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123
  Male | 174
Region of Enrollment [Number; unit: participants]
  United States | 297

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number of participants with Adverse Events
Time Frame: 5 Years
Measure: Number; unit: participants
Groups:
- Implanted With Biocor, Biocor Supra, Biocor Mitral Valves: Biocor (aortic), Biocor Supra (aortic) and Biocor Mitral valves: Replacement for a diseased, damaged, malformed aortic or mitral heart valve
Arm/Group | Implanted With Biocor, Biocor Supra, Biocor Mitral Valves
Number analyzed (Participants) | 297
participants
  Mortality-valve related | 6
  Mortality-cardiac related | 14
  Bleed | 53
  Embolism | 10
  Endocarditis | 10
  Reoperation-explant | 13
  Structural Deterioration | 3
  Thrombosis | 1

2. Primary Outcome: Characterize Patient NYHA Functional Classification Status
Description: The New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life.
  Class I. Patients with cardiac disease but without resulting limitation of physical activity.
  Class II. Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest.
  Class III. Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest.
  Class IV. Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest.
  The Criteria Committee of the New York Heart Association. Nomenclature and Criteria for Diagnosis of Diseases of the Heart and Great Vessels. 9th ed. Boston, Mass: Little, Brown & Co; 1994:253-256.
Time Frame: 5 year
Population: Number of participants that completed the visit and assessment
Measure: Number; unit: participants
Arm/Group | Implanted With Biocor or Biocor Supra Valves
Number analyzed (Participants) | 106
participants
  NYHA I | 73
  NYHA II | 24
  NYHA III | 9
  NYHA IV | 0

3. Primary Outcome: Characterize the Hemodynamic Performance of the Valve
Description: Gradient is the pressure difference from one side of the valve to the other side of the valve. For this study pressure is measured in mmHg.
  Mean gradient for each patient is the average of the pressure differences from one side of the valve to the other side of the valve.
Time Frame: 5 Year
Population: Number of participants that completed the visit and assessment
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Biocor Valve: Biocor valves: Replacement for a diseased, damaged, malformed aortic heart valve
Arm/Group | Biocor Valve | Biocor Supra Valve | Biocor Mitral Valve
Number analyzed (Participants) | 43 | 30 | 17
mmHg
  19mm | NA (NA) — no subjects implanted with this size valve followed through 5 years | 17.8 (7.8) | NA (NA) — no subjects implanted with this size valve followed through 5 years
  21mm | 20.5 (8.1) | 12.7 (5.9) | NA (NA) — no subjects implanted with this size valve followed through 5 years
  23mm | 16.7 (6.3) | 15.1 (4.9) | NA (NA) — no subjects implanted with this size valve followed through 5 years
  25mm | 11.3 (5.5) | 9.0 (2.3) | NA (NA) — no subjects implanted with this size valve followed through 5 years
  27mm | 14.4 (4) | 5.6 (0) | 4.2 (0.6)
  29mm | 11.3 (7.3) | NA (NA) — no subjects implanted with this size valve followed through 5 years | 3.7 (2.3)
  31mm | NA (NA) — no subjects implanted with this size valve followed through 5 years | NA (NA) — no subjects implanted with this size valve followed through 5 years | 1.9 (0.7)
  33mm | NA (NA) — no subjects implanted with this size valve followed through 5 years | NA (NA) — no subjects implanted with this size valve followed through 5 years | 2.0 (0.8)

ADVERSE EVENTS:
Arm/Group | Implanted With Biocor or Biocor Supra Valves
Serious Adverse Events (participants affected / at risk) | 91/297
Other Adverse Events (participants affected / at risk) | 0/297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Implanted With Biocor or Biocor Supra Valves (N=297)
Major Bleed (Vascular disorders) | 50
Minor Bleed (Vascular disorders) | 4
Embolism (Nervous system disorders) | 10
Endocarditis (Cardiac disorders) | 10
Reoperation-Explant (Surgical and medical procedures) | 13
Structural Deterioration (Cardiac disorders) | 3
Thrombosis (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other